CLINICAL TRIAL: NCT02782364
Title: Evaluation of the Fast Fill Technique for Anal Acoustic Reflectometry (AAR) in the Incontinent Anal Sphincter
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2015GA004
Record Dates: First submitted 2016-05-12; First posted 2016-05-25 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Faecal Incontinence
Keywords: Faecal Incontinence
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Faecal Incontinence: fast-fill measurement first: Observational study where patients with faecal incontinence undergo two AAR measurements; one with the original step-wise technique and the second with the newer fast-fill technique. A further standard manometry measurement will be taken. 18 patients will undergo fast-fill measurement first.
- Faecal Incontinence: step-wise measurement first.: Observational study where patients with faecal incontinence undergo two AAR measurements; one with the original step-wise technique and the second with the newer fast-fill technique. A further standard manometry measurement will be taken. 18 patients will have step-wise measurement first.

SUMMARY:
Anal Acoustic Reflectometry (AAR) is a technique that has been studied in our department over the last 6 years. Sound waves pass into a balloon placed in the anal canal and are used to measure the cross-sectional area. By gradually increasing and decreasing the pressure in the balloon the investigators can measure the pressure at which the cross-sectional area starts to increase and decrease, and the anal canal starts to open and close. This assessment mimics the natural opening and closing of the anal canal and the effect of squeezing the muscles.

The gold standard investigation of the anal sphincter muscles has been manometry which measures anal canal pressure at rest and during squeeze. However, it has limitations. Despite the two measurements being within the normal range, some patients can have significant faecal incontinence. This has prompted clinicians to search for a better investigation to guide the management of this condition.

AAR is a reproducible and repeatable technique that has been used as a research technique in the assessment of faecal incontinence. It has been shown to correlate with symptom severity and, unlike manometry, is able to distinguish between different symptomatic subgroups with faceal incontinence. In our studies so far the investigators have increased the bag inflation pressure a step at a time which means that each study takes about 20 minutes to perform. The limitation of this method is that during the measurement of squeeze pressure the sphincter muscle is subject to fatigue. A recent study using the acoustic technique in the urethra has demonstrated a faster method of recording measurements over an 8 minute period. The investigators propose to study the fatiguability effects of this faster technique and validate the method against the existing step-wise technique and standard anal manometry.

Patients will be randomised into two groups:

1. Stepwise then fast-fill
2. Fast-fill then stepwise

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years
* have capacity to consent to the study
* patients with symptoms of faecal incontinence

Exclusion Criteria:

* minors under age of 18 years old
* patients who lack capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the pelvic floor clinic and neurogastroenterology with symptoms of faecal incontinence
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Telford, MBChBMDFRCS, Study Chair — University Hospital of South Manchester
Locations (1):
- University Hospital of South Manchester, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
individual patient data will not add any further information to the overall data

REFERENCES:
- [Background] Klarskov N, Saaby ML, Lose G. A faster urethral pressure reflectometry technique for evaluating the squeezing function. Scand J Urol. 2013 Dec;47(6):529-33. doi: 10.3109/21681805.2013.776629. Epub 2013 Mar 19. PMID 23506115
- [Background] Hornung BR, Mitchell PJ, Carlson GL, Klarskov N, Lose G, Kiff ES. Comparative study of anal acoustic reflectometry and anal manometry in the assessment of faecal incontinence. Br J Surg. 2012 Dec;99(12):1718-24. doi: 10.1002/bjs.8943. PMID 23132420
- [Background] Klarskov N. Urethral pressure reflectometry. A method for simultaneous measurements of pressure and cross-sectional area in the female urethra. Dan Med J. 2012 Mar;59(3):B4412. PMID 22381095
- [Background] Mitchell PJ, Klarskov N, Telford KJ, Hosker GL, Lose G, Kiff ES. Viscoelastic assessment of anal canal function using acoustic reflectometry: a clinically useful technique. Dis Colon Rectum. 2012 Feb;55(2):211-7. doi: 10.1097/DCR.0b013e31823b2499. PMID 22228166
- [Background] Mitchell PJ, Klarskov N, Telford KJ, Hosker GL, Lose G, Kiff ES. Anal acoustic reflectometry: a new reproducible technique providing physiological assessment of anal sphincter function. Dis Colon Rectum. 2011 Sep;54(9):1122-8. doi: 10.1097/DCR.0b013e318223fbcb. PMID 21825892
- [Background] Saaby ML, Klarskov N, Lose G. Urethral pressure reflectometry before and after tension-free vaginal tape. Neurourol Urodyn. 2012 Nov;31(8):1231-5. doi: 10.1002/nau.22239. Epub 2012 Mar 27. PMID 22457059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients attending clinic for routine evaluation of faecal incontinence were approached to particpate in this study
Groups:
- Stepwise First, Then Fast-fill: Observational study where patients with faecal incontinence undergo two AAR measurements; one with the original step-wise technique and the second with the newer fast-fill technique. A further standard manometry measurement will be taken. To reduce the bias of one test on the other, the order of the test were randomised so that half of the patients will undergo stepwise measurement first and another half of the patients will have stepwise measurement first. Patients in this arm underwent stepwise, followed by a two minute rest, then fast fill, followed by a two minute rest, and then by manometry
- Fast-fill First, Then Stepwise: Observational study where patients with faecal incontinence undergo two AAR measurements; one with the original step-wise technique and the second with the newer fast-fill technique. A further standard manometry measurement will be taken. To reduce the bias of one test on the other, the order of the test were randomised so that half of the patients will undergo fast-fill measurement first and another half of the patients will have step-wise measurement first. Patient min this arm underwent fast fill, followed by a two minute rest, then step wise, followed by a two minute rest, and then by manometry
Period: Overall Study
Arm/Group | Stepwise First, Then Fast-fill | Fast-fill First, Then Stepwise
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis of a total of 32 patients was performed. Measurement data from four patients was not able to be accurately interpreted
Groups:
- Faecal Incontinence: Observational study where patients with faecal incontinence undergo two AAR measurements; one with the original step-wise technique and the second with the newer fast-fill technique. A further standard manometry measurement will be taken. 16 patients will undergo fast-fill measurement first and another 16 patients will have step-wise measurement first
Arm/Group | Faecal Incontinence
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants] — Population: Analysis of a total of 32 patients was performed. Measurement data from four patients was not able to be accurately interpreted
  Participants
    <=18 years | 0
    Between 18 and 65 years | 23
    >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 60 [32 to 75]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measurement data from four patients was not able to be accurately interpreted
  Participants
    Female | 26
    Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: Measurement data from four patients was not able to be accurately interpreted
  participants
    United Kingdom | 32

OUTCOME MEASURES:

1. Primary Outcome: Opening Pressure
Description: Opening Pressure (Op - cm H2O) - the point at which the anal canal just begins to open
Time Frame: 10 minutes
Measure: Median (Full Range); unit: cmH2O
Groups:
- Stepwise; Fast-fill: Observational study where patients with faecal incontinence undergo two AAR measurements; one with the original step-wise technique and the second with the newer fast-fill technique.
Arm/Group | Stepwise | Fast-fill
Number analyzed (Participants) | 32 | 32
cmH2O | 35.13 [9.87 to 102.7] | 37.5 [13.84 to 117.7]

2. Primary Outcome: Opening Elastance
Description: Opening Elastance (Oe - cm H2O/mm2) - the resistance of the anal canal to stretch
Time Frame: 10 minutes
Measure: Median (Full Range); unit: cm H2O/mm2
Arm/Group | Stepwise | Fast-fill
Number analyzed (Participants) | 32 | 32
cm H2O/mm2 | 0.84 [0.7 to 1.04] | 1.31 [0.7 to 2.41]

3. Primary Outcome: Closing Pressure
Description: Closing Pressure (Cp - cm H2O) - the pressure at which the anal canal closes after a period of opening
Time Frame: 10 minutes
Measure: Median (Full Range); unit: cmH2O
Arm/Group | Stepwise | Fast-fill
Number analyzed (Participants) | 32 | 32
cmH2O | 27.22 [7.97 to 97.44] | 22.7 [5.35 to 82.35]

4. Primary Outcome: Closing Elastance
Description: Closing Elastance (Ce - cm H2O/mm2) - the ability of the anal canal to close passively after a period of stretch
Time Frame: 10 minutes
Measure: Median (Full Range); unit: cm H2O/mm2
Arm/Group | Stepwise | Fast-fill
Number analyzed (Participants) | 32 | 32
cm H2O/mm2 | 0.88 [0.41 to 1.57] | 1.11 [0.58 to 2.07]

5. Primary Outcome: Hysteresis
Description: Hysteresis (%) - the energy dissipated during opeing and closing of the anal canal
Time Frame: 10 minutes
Measure: Median (Full Range); unit: percentage
Arm/Group | Stepwise | Fast-fill
Number analyzed (Participants) | 32 | 32
percentage | 19.04 [1.62 to 53.01] | 35.75 [20.33 to 52.57]

6. Primary Outcome: Squeeze Opening Pressure
Description: Squeeze opening pressure (SqOp - cm H20) - the pressure at which the anal canal just starts to open whilst the patient is voluntarily trying to keep the anal canal closed
Time Frame: 10 minutes
Measure: Median (Full Range); unit: cmH2O
Arm/Group | Stepwise | Fast-fill
Number analyzed (Participants) | 32 | 32
cmH2O | 59.47 [9.15 to 200] | 69.87 [19.65 to 156]

7. Primary Outcome: Squeeze Opening Elastance
Description: Squeeze opening elastance (Sq)e - cm H20/mm2) - the resistance of the anal canal to stretch whilst the patient is voluntarily trying to keep the anal canal closed
Time Frame: 10 minutes
Measure: Median (Full Range); unit: cmH20/mm2
Arm/Group | Stepwise | Fast-fill
Number analyzed (Participants) | 32 | 32
cmH20/mm2 | 1.06 [0.44 to 2.6] | 1.27 [0.87 to 2.2]

8. Secondary Outcome: Manometry - Resting Pressure
Description: anal manometry measured in cmH20
Time Frame: 10 minutes
Population: 29 patient analysed due to equipment issues performing for other 3 patients. It was pre-specified to combine data collected from the manometry regardless of the sequence of administration of techniques for AAR measurements as previous study had previously shown that the order of data collection did not impact on the measurements obtained
Measure: Median (Full Range); unit: cmH20
Groups:
- Faecal Incontinence: Observational study where patients with faecal incontinence undergo two AAR measurements; one with the original step-wise technique and the second with the newer fast-fill technique. A further standard manometry measurement will be taken. 18 patients will undergo fast-fill measurement first and another 18 patients will have step-wise measurement first.
  This study is classed as observational as the randomisation is solely the order in which the two tests are performed. The test itself can be performed at can be performed at different rates and this study is to evaluate the two
Arm/Group | Faecal Incontinence
Number analyzed (Participants) | 29
cmH20 | 45 [15 to 151]

ADVERSE EVENTS:
Time Frame: Patients were recruited over a 12 month window. This study treatment and data was collected on one day (a point in time measurement) and any adverse events (if present) would occur at the time of measurement. If no events were noted at this point, then further data was not collected
Description: AEs or SAEs would occur during or directly after the procedure and noted by the attending clinician.
Groups:
- Stepwise First, Then Fast-fill: Stepwise First, Then Fast-fill measurement. Observational study where patients with faecal incontinence undergo two AAR measurements; first with the original step-wise technique and the second with the newer fast-fill technique. A further standard manometry measurement will be taken. To reduce the bias of one test on the other, the order of the test were randomised so that half of the patients will undergo stepwise measurement first and another half of the patients will have stepwise measurement first. Patients in this arm underwent stepwise, followed by a two minute rest, then fast fill, followed by a two minute rest, and then by manometry
  Previous Work has been carried out looking at the sequence has shown no difference in the order. Therefore to keep consistency this method has been continued and results combined
- Fast-fill First, Then Stepwise: Fast-fill measurement then Stepwise measurement. Observational study where patients with faecal incontinence undergo two AAR measurements; with the newer fast-fill technique and the second with the original step-wise technique. A further standard manometry measurement will be taken. To reduce the bias of one test on the other, the order of the test were randomised so that half of the patients will undergo fast-fill measurement first and another half of the patients will have step-wise measurement first. Patient min this arm underwent fast fill, followed by a two minute rest, then step wise, followed by a two minute rest, and then by manometry.
  Previous Work has been carried out looking at the sequence has shown no difference in the order. Therefore to keep consistency this method has been continued and results combined
Arm/Group | Stepwise First, Then Fast-fill | Fast-fill First, Then Stepwise
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes